CLINICAL TRIAL: NCT05297435
Title: Psychotraumatology in Somatic Medicine - Gynecological Consultation
Brief Title: Psychotraumatology in Somatic Medicine
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Katja Haemmerli Keller, Dr. phil., Cantonal Hospital of St. Gallen
Other Study IDs: 2020-02551
Record Dates: First submitted 2022-03-11; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Trauma, Psychological; Somatic
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaires — Questionnaire study

SUMMARY:
Psychotraumatology is clinically highly relevant, especially in the medical-somatic disciplines. Despite progress in recent decades, the clinical care is still inadequate - with unfavorable health effects for affected patients. There are avoidable burdens for involved clinicians and the health care system as a whole, also in terms of costs. With this background, our long-term project combines different research levels. Besides clarifying the clinical phenomenon, it aims to examine 1) the influence of traumatization on the physician-patient interaction as well as 2) the current psychological stress of the patients. Furthermore, 3) moderating factors on the side of the physicians, such as professional experience on the physician-patient interaction will be examined.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Female patients of the preventive consultation of the gynecological clinic of the cantonal hospital St.Gallen

Exclusion Criteria:

* Severe mental disorder (e.g. dissociative disorder)
* Insufficient knowledge of German

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients of the preventive consultation of the gynecological clinic of the cantonal hospital St.Gallen
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of physician-patient relationship | Day 0
  German version of the questionnaire "Patient Reactions Assessment Instruments" (PRA-D; Brenk-Franz et al., 2016)

SECONDARY OUTCOMES:
Early traumatization | Day 0
  German version of the questionnaire "Childhood Trauma Questionnaire" (CTQ, Bernstein und Fink, 1998)
Current traumatization | Day 0
  German version of the questionnaire "Impact of Event Scale-Revised" (IES-R; Weiss & Marmar, 1997)
Anxiety & Depression | Day 0
  German version of the questionnaire "Hospital Anxiety and Depression Scale" (HADS; Herrmann et al., 1995; Hermann-Lingen et al., 2011)
Dissociative symptoms | Day 0
  German questionnaire on dissociative symptoms (FDS-20; Spitzer et al., 2021)
General distress | Day 0
  German version of the questionnaire "distress thermometer" (BTH; Mehnert et al., 2006)

CONTACTS AND LOCATIONS:
Locations (1):
- Katja Haemmerli Keller, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No